CLINICAL TRIAL: NCT04248751
Title: A Prospective, Randomized Evaluation of Bioinductive Augmentation for High Risk Rotator Cuff Tears
Brief Title: Evaluating the Use of a Bioinductive Graft in Treating Massive Rotator Cuff Tears
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ivan Wong (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ivan Wong, MD Orthopedic Surgeon, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Regen
Record Dates: First submitted 2019-11-15; First posted 2020-01-30 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Rotator Cuff Tear; Rotator Cuff Injury
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Debridement

STUDY DESIGN:
Intervention Model Description: Patients that have consented to the study will be randomized into 2 groups with a 50% chance of being in either group. Patients will be blinded and assessed by blinded assessors. Only after the one-year mark will the patient become unblinded following being asked which intervention they believe they received.
  Crossover design: Among those 38 patients without augmentation, we anticipate that 23 of them will have re-tear (assuming a 60% re-tear rate). We will offer them revision surgery with augmentation. Then those patients will be followed up 1 year and 2-years afterwards. MRI follow-up will be done at 1 year postoperatively to assess the healing rates. Outcome scores (as per above) will be collected at each follow-up and compared with their non-augmented scores to assess the improvement.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graft-Augmented (Experimental): Patients randomized to this group will receive a regular rotator cuff repair where the bursa will be debrided thoroughly, and rotator cuff edges will be shaved down to stable tissue. The rotator cuff will be repaired using multiple single row triple loaded suture anchor placed adjacent to the articular margin. Then, the graft will be delivered to the subacromial space and positioned over the bursal surface of the suprasinatus tendon, ensuring that the lateral edge of the implant will overlap with the head of the humerus. The graft will be fixed with tendon and bone staples.
  Interventions: Device: Regeneten
- Non-augmented (Active Comparator): Patients randomized to this group will receive a regular rotator cuff repair where the bursa will be debrided thoroughly, and rotator cuff edges will be shaved down to stable tissue. The rotator cuff will be repaired using multiple single row triple loaded suture anchor placed adjacent to the articular margin.
  Interventions: Procedure: Debridement

INTERVENTIONS:
Device: Regeneten — A new scaffold material made of highly purified, type I collagen from bovine tendons has shown great promise as a bioinductive implant that helps induce the formation of new tendon-like tissue over the surface of partial- or full-thickness rotator cuff tears. This new graft material has the benefit of decreasing surgery time, as it takes a few minutes to put in place, while increasing healing and tendon thickness.
  Arms: Graft-Augmented
Procedure: Debridement — The bursa will be debrided thoroughly, and rotator cuff edges will be shaved down to stable tissue. The rotator cuff will be repaired using multiple single row triple loaded suture anchor placed adjacent to the articular margin
  Arms: Non-augmented

SUMMARY:
The rotator cuff is a complex of 4 tendons that aid in stabilizing and moving the shoulder. Rotator cuff tears are common shoulder injuries in adults. While some tears can be managed by physiotherapy, other rotator cuff tears will require surgery. On occasion, when a person has had a large rotator cuff tear for a long period of time, the tear can grow and the tendons retract. This effect makes it very difficult for the tendons to be repaired to their normal spot.

The most common surgical technique employed to manage a tear that cannot be repaired is to remove all unhealthy, inflamed scar tissue in a process called debridement. Often there is a bone spur that must be shaved down as well. This can help to reduce the pain in the patient as well as assist the range of motion slightly but will not prevent the tear becoming larger. This will also not prevent a re-tear of the tendons.

Recently, surgeons have begun using a variety of materials to help reconstruct torn rotator cuffs. New grafts made of highly purified collagen from bovine tendons has been used to bridge large gaps in the tendons, and repair the tendon back to the bone. This technique has been done many times by skilled shoulder surgeons in Canada, the United States and around the world.

Initial reports by surgeons who do this procedure show that the patients have less pain and better range of motion than before the surgery. Shoulder surgeons do not know which is the better treatment for large rotator cuff tears. Both treatments (graft and debridement) can reduce pain and improve movement of the shoulder. The purpose of this study is to help determine whether patients who receive an allograft have better function and fewer re-tear at one year after surgery than those who received a debridement alone.

DETAILED DESCRIPTION:
Rotator cuff injuries are among the most common soft tissue injuries of the shoulder. Characterized by insidious onset of progressive pain and weakness, with concomitant loss of range of motion, patients with pathological conditions of the rotator cuff are often unable to associate the onset of symptoms with a specific traumatic event. Loss of continuity of the rotator cuff can be described in several ways, including acute or chronic, partial or full-thickness and traumatic or degenerative. For this study, only patients with radiography confirmed large rotator cuff tears (> 3 cm) resulting from trauma and/or degeneration will be observed.

Historically, many operative procedures have been used by surgeons in the treatment of large rotator cuff tears including open rotator cuff repair, mini- open rotator cuff repair, arthroscopic rotator cuff repair, bridging techniques, debridement, arthroscopic rotator cuff repair with acromioplasty, arthroscopic rotator cuff repair without acromioplasty, surgical augmentation, debridement etc. While the surgical repair of large rotator cuff tears has resulted in pain relief and improved function, the re-tear rate (55%-94%) has remained high despite advances in repair techniques. The re-tear rates correlate with the size of the rotator cuff tear as well as with other factors such as muscle atrophy, tendon quality, and postoperative rehabilitation protocol.

With an effort to improve healing rates, surgeons have used various biologic tissues to either substitute for or augment the repair of the rotator cuff. These tissues include the patients' biceps tendon, fascia latae allografts and autografts, freeze-dried rotator cuff allografts, and synthetic materials such as polypropylene mesh.1 A new scaffold material made of highly purified, type I collagen from bovine tendons has shown great promise as a bioinductive implant that helps induce the formation of new tendon-like tissue over the surface of partial- or full-thickness rotator cuff tears.This new graft material has the benefit of decreasing surgery time, as it takes a few minutes to put in place, while increasing healing and tendon thickness.

The investigators hypothesize that arthroscopic augmentation using a bioinductive collagen implant will have superior outcomes in terms of increasing healing, thereby decreasing re-tear rate, as compared to participants who are treated with the current gold standard treatment (consisting of debridement, acromioplasty, and rotator cuff repair). The investigators hypothesize that the participants with graft augment will have decreased pain both during the early recovery phase and two years post-operatively as compared to the non-augmented group. Additionally, the investigators hypothesize that participants with the collagen scaffold will have better outcome scores at two years, as compared to the non-augmented group.

ELIGIBILITY:
Inclusion Criteria:

* Magnetic resonance imaging (MRI) proven diagnosis of a large >3cm tear of the shoulder rotator cuff in a competent adult (>18 years of age).

Exclusion Criteria:

* Patients with subscapular tear
* Glenohumeral osteoarthritis
* A normalized WORC score >70 (where scores range between 0-100, and 100 is the best outcome)
* Uncontrolled diabetes (Hgb A1C >7%)
* Pregnancy
* Presence of local or systemic infection
* Inability to cooperate with and/or comprehend post-operative instructions
* Nonvascular surgical sites (MRI proven)
* Poor nutritional state (Alb <30 g/L)
* Cancer
* Paralysis of the shoulder
* Contracture of the shoulder
* Presence of cuff tear arthropathy or osteoarthritis of the shoulder
* Patients unable to provide informed consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Healing | 2 years
  A change in healing to be assessed by comparing re-tear rates.

SECONDARY OUTCOMES:
VAS Pain | Early recovery phase and 2 years
  Pain will be assessed using the Visual Analogue Scale (VAS) pain scale, a scale from 1 to 10 where 10 represents the best health and 1 represents worse health.
Western Ontario Rotator Cuff Index | 1 and 2 years
  A questionnaire used to determine shoulder function in patients with rotator cuff tears
Marx Shoulder Activity Scale | 1 and 2 years
  Activity survey that is short, easy to administer and is a good measure of shoulder activity which could be used to predict outcome of shoulder disorders
Disabilities of the Arm Shoulder and Hand (DASH) Questionnaire | 1 and 2 years
  The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms.
American Shoulder and Elbow Surgeons (ASES) Questionnaire | 1 and 2 years
  American Shoulder and Elbow Surgeons (ASES) questionnaire is a validated, self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms.
Veterans Rand 12-Item Health Survey (VR12) | 1 and 2 years
  Questionnaire used to assess general health
EQ5D-5L | 1 and 2 years
  Questionnaires used to assess general health that is also commonly used during economic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Wong, MD, Principal Investigator — Orthopaedic Surgeon
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No